CLINICAL TRIAL: NCT05288257
Title: The Role Cognitive Non-technical Skills Learning Module in Promoting A Safe Laparoscopic Cholecystectomy: Critical Analysis on Situation Awareness and Intraoperative Decision Making in the Prevention of Complications
Brief Title: Mixed Method Study Protocol_Cognitive Non-technical Skills Learning Module for a Safe Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RSUP Fatmawati (Other)
Responsible Party: Principal Investigator, Adianto Nugroho, Principal Investigator, RSUP Fatmawati
Other Study IDs: 22-01-0029
Record Dates: First submitted 2022-02-08; First posted 2022-03-21 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Learning Module; Cognitive Non-technical Skills
Keywords: Safe Laparoscopic Cholecystectomy; Situation Awareness; Decision Making

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Learning Module — Safe Cholecystectomy Learning Module
  Other Names: Safe Cholecystectomy

SUMMARY:
A mixed-methods sequential explanatory design study. The first quantitative phase will be an online survey to surgeons that includes questions related to their experience learning and performing laparoscopic cholecystectomy. The second qualitative phase will use depth interview to elaborate surgeon's experience regarding a safe laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Bile duct injuries from laparoscopic cholecystectomy remain a significant source of morbidity and are often the result of intraoperative errors in perception, judgment, and decision-making. Cognitive non-technical skills namely situation awareness and decision-making skills are essential in doing a safe laparoscopic cholecystectomy, as in any kind of surgery. Studies regarding cognitive non-technical skills and how to teach them are still lacking, especially in the field of surgery.

With this study, the investigators aim to formulate a comprehensive learning module for a safe laparoscopic cholecystectomy accomodating cognitive non-technical skills based on the surgeon's experience while learning and doing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons and / or surgical residents
* Complete all the required documents

Exclusion Criteria:

* Refuse to participate in one or more parts of the study

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgeons and Surgical residents
Sampling Method: Non-Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative: Community Survey | February - March 2022
  Survey data
Qualitative: In Depth Interview | March - April 2022
  Semi-structured interview data obtained from In Depth Interview
Qualitative: Delphi Study | May 2022
  Learning Module

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Fatmawati, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No